CLINICAL TRIAL: NCT07089498
Title: 13C-Octanoic Acid Breath Test for the Evaluation of a Low-fodmaps Diet on Gastric Emptying in Celiac Patients With Functional Disorders
Brief Title: 13C-Octanoic Acid Breath Test on Gastric Emptying in Celiac Patients With Functional Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2557
Record Dates: First submitted 2023-01-04; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2022-12

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Fodmap Gluten Free Diet (Experimental): Patients received dietary advice in the form of a table divided into two columns, one reporting the allowed food because low in FODMAPs and the other indicating the prohibited food due to its high continent of FODMAPs
  Interventions: Other: Dietary Intervention (Low Fodmap Gluten Free Diet)
- Regular Gluten Free Diet (No Intervention): Patients received a table containing a list of allowed food based on a regular diet

INTERVENTIONS:
Other: Dietary Intervention (Low Fodmap Gluten Free Diet) — The intervention provides the administration of a Low Fodmap Diet to celiac or non celiac patients with functional gastrointestinal disorders
  Arms: Low Fodmap Gluten Free Diet

SUMMARY:
The goal of this interventional study is the evaluation of a diet low in fodmaps on gastric emptying in celiac patients with functional disorders.

DETAILED DESCRIPTION:
The goal of this interventional study is the evaluation of a diet low in fodmaps on gastric emptying in celiac patients with functional disorders.

The aims of the study are:

* Evaluation of gastric emptying time by a 13C-Octanoic Acid Breath Test, pre and post-diet (T1 and T2) in celiac patients with functional dyspepsia and non-celiac patients with functional dyspepsia.
* Evaluation of gastrointestinal symptoms, quality of life, and mental health in patients with non-celiac and celiac functional disorders pre- and post-diet (T1 and T2).

Participants:

* Will run the 13C-octanoic acid breath test pre- and post-diet
* Will complete the VAS, SF-36, and SCL-90 questionnaires pre- and post-diet
* Will follow a low fodmap gluten free diet or a regular gluten-free diet for six weeks Researchers will compare celiac and non-celiac patients.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥ 18 years old
* gender: male or female
* patients who have signed informed consent
* patients diagnosed with a functional gastrointestinal disorder who meet Rome IV criteria (according to Rome Foundation's latest revision of 2016)

Exclusion Criteria:

* patients who have not given informed consent
* patients without a diagnosis of a functional gastrointestinal disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluating gastric emptying time by a 13C-Octanoic Acid Breath Test, pre and post-diet (T1 and T2) in celiac patients with functional dyspepsia and non-celiac patients with functional dyspepsia | Six weeks
  Evaluating gastric emptying time by a 13C-Octanoic Acid Breath Test, pre and post-diet

SECONDARY OUTCOMES:
Comparison of the effects of dietary recommendation for a diet low in Oligo-, Di- and Monosaccharides and Polyols (FODMAPs) or a balanced diet in celiac and non-celiac dyspeptic patients on gastric emptying time | Six weeks
  Comparison of the effects of dietary recommendation for a diet low in Oligo-, Di- and Monosaccharides and Polyols (FODMAPs) or a balanced diet in celiac and non-celiac dyspeptic patients on gastric emptying time
Evaluation of gastrointestinal symptoms (VAS) | Six weeks
  Evaluation of gastrointestinal symptoms through Visual Analogue Scale (VAS) in celiac and non-celiac dyspeptic patients pre- and post-nutritional intervention (t1 and t2)
Evaluation of quality of life (SF-36) | Six weeks
  Evaluation of quality of life through a questionnaire on the health state (Short Form Health Survey, SF-36) in celiac and non-celiac dyspeptic patients pre- and post-nutritional intervention (t1 and t2)
Evaluation of mental health (SCL-90) | Six weeks
  Evaluation of mental health through a questionnaire on the health state (Symptom Check List, SCL-90) in celiac and non-celiac dyspeptic patients pre- and post-nutritional intervention (t1 and t2)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Elli, PhD, MD, Principal Investigator — IRCCS Maggiore H
Locations (2):
- Italy (2):
  - Leda Roncoroni, Milan
  - Luca Elli, Milan

REFERENCES:
- [Background] Bruno G, Lopetuso LR, Ianiro G, Laterza L, Gerardi V, Petito V, Poscia A, Gasbarrini A, Ojetti V, Scaldaferri F. 13C-octanoic acid breath test to study gastric emptying time. Eur Rev Med Pharmacol Sci. 2013;17 Suppl 2:59-64. PMID 24443070
- [Background] Usai Satta P, Scarpa M, Oppia F, Loriga F. 13C-octanoic acid breath test in functional and organic disease: critical review of literature. Eur Rev Med Pharmacol Sci. 2005 Sep-Oct;9(5 Suppl 1):9-13. PMID 16457124
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Prunas A, Sarno I, Preti E, Madeddu F, Perugini M. Psychometric properties of the Italian version of the SCL-90-R: a study on a large community sample. Eur Psychiatry. 2012 Nov;27(8):591-7. doi: 10.1016/j.eurpsy.2010.12.006. Epub 2011 Feb 21. PMID 21334861
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Massironi S, Branchi F, Fraquelli M, Baccarin A, Somalvico F, Ferretti F, Conte D, Elli L. Effects of a Gluten-Containing Meal on Gastric Emptying and Gallbladder Contraction. Nutrients. 2018 Jul 16;10(7):910. doi: 10.3390/nu10070910. PMID 30012987